CLINICAL TRIAL: NCT03165682
Title: Fatigue, Depression, and Cortical Excitability Changes in Systemic Lupus Erythematosus
Brief Title: Fatigue, Depression, and Cortical Excitability in Systemic Lupus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mary Jacob Ross, Principal investigator, Assiut University
Other Study IDs: FDCS
Record Dates: First submitted 2017-05-20; First posted 2017-05-24 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Systemic Lupus Erythematosus
Keywords: fatigue; depression; cortical excitability
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Fatigue; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Twenty-five patients with Systemic Lupus Erythematosus with prominent fatigue symptoms ( inclusion criterion: FSS of at least 4)
- Group 2: Twenty-five patients with Systemic Lupus Erythematosus without subjectively enhanced fatiguability
- Group 3: Twenty-five age, sex and educationally matched controls among the health worker.

SUMMARY:
Systemic lupus erythematosus is a chronic inflammatory autoimmune disease with an unknown cause and many challenges. Whilst corticosteroids and effective immunosuppressive therapy have transformed the management of patients with active systemic lupus erythematosus, one of the major causes of morbidity in Systemic lupus erythematosus patients is chronic, debilitating fatigue.

Despite frequent occurrence of fatigue in Systemic Lupus Erythematosus, to the best of our knowledge, no studies have been directly performed to examine fatigue-related changes in cortical motor function in Systemic lupus erythematosus. In this study, we hypothesized that Systemic lupus erythematosus patients with fatigue and depression versus Systemic lupus erythematosus patients without fatigue and depression would present an alteration of motor cortex excitability.

DETAILED DESCRIPTION:
Fatigue, is a multidimensional phenomenon that affects individuals physically, emotionally, cognitively, and behaviorally.It affects 80-90% of patients with systemic lupus erythematosus. It is likely multifactorial and may be caused by disordered sleep, anxiety and depression, pain, polypharmacy, comorbidities, and possibly disease activity.

Additionally, fatigue is the most prevalent symptom in systemic lupus erythematosus, being present in up to 90% of patients. Moreover, fatigue has a major impact on the Health-Related Quality Of Life of Systemic lupus erythematosus patients through its impact on family life, work, social life, emotional wellbeing, and cognition. Therefore, every effort should be made to relieve fatigue in this population. Recommendations for the management of fatigue usually combine pharmacologic and nonpharmacologic interventions; however, no speciﬁc drugs have proven useful for treating fatigue in Systemic lupus erythematosus.

ELIGIBILITY:
Inclusion Criteria:

* All the participants:

  1. 18 years of age or older.
  2. For Systemic lupus patients: have a stable drug regimen for 3 months prior to study entry; disease duration for at least 6 months or longer
  3. able to give written consent for participation.
  4. able to understand and respond the questionnaires.
  5. be free of serious comorbid medical conditions such as diabetes, congestive heart failure, renal failure, cancer, or fibromyalgia, which would confound interpretations of health status; and not pregnant.

Exclusion Criteria:

* Any patient will meet any of these conditions will be excluded from the study, that including:

  1. Patient less than 18 years old.
  2. Patients with a definite diagnosis of any other systemic autoimmune disorders.
  3. History of any other neurologic disease, seizure or major medical disorders including heart failure, respiratory compromise, renal insufficiency, hepatic dysfunction, diabetes mellitus, malignancy, or endocrinal disturbance.
  4. Other contraindications of Transcranial Magnetic Stimulation as:

     1. Personal or family history of epilepsy, brain tumor, brain injury.
     2. History of metallic particles in the eye or head outside the mouth,
     3. Cardiac pacemakers, implanted neurostimulators, cochlear implants, implanted medication pumps.
     4. History of drug or alcohol abuse.
     5. Pregnancy.
     6. Comedication with neuroleptics and tricyclic antidepressants (amitriptyline etc.)
     7. Patients with increased intracranial pressure (which lowers seizure threshold intracardiac line).
     8. Significant heart disease: extensive ischemia.
     9. Bipolar disorder.
     10. History of stroke or other brain lesions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: not related
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Cortical excitability assessment among studied participants. | six months
  Done by Transcranial Magnetic Stimulation :
  For assessment of cortical excitability parameters (resting and active motor threshold Cortical Silent Period at different intensities) among studied participants.

SECONDARY OUTCOMES:
Depression assessment among studied participants. | six months
  The Beck Depression Inventory (BDI), self-assessment question, is one of the most widely used instruments to evaluate the severity of depression. The results were evaluated by a psychiatrist.

CONTACTS AND LOCATIONS:
Overall Officials: Rania M. Gamal-El Din, Assistant Professor Dr, Study Director — Assiut University; Eman M. El-Hakeem, Lecturer Dr, Study Director — Assiut University

REFERENCES:
- [Result] Li J, May W, McMurray RW. Pituitary hormones and systemic lupus erythematosus. Arthritis Rheum. 2005 Dec;52(12):3701-12. doi: 10.1002/art.21436. No abstract available. PMID 16320320
- [Result] McMurray RW, May W. Sex hormones and systemic lupus erythematosus: review and meta-analysis. Arthritis Rheum. 2003 Aug;48(8):2100-10. doi: 10.1002/art.11105. No abstract available. PMID 12905462